CLINICAL TRIAL: NCT03387306
Title: Reduced Serum Bilirubin Levels in Patients With Normal-tension Glaucoma
Brief Title: Serum Bilirubin Levels in Normal-tension Glaucoma
Status: Completed | Type: Observational
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Sadık Altan Ozal, Assistant of Proffessor, Trakya University
Other Study IDs: 14783786
Record Dates: First submitted 2017-12-21; First posted 2018-01-02 (Actual); Last update posted 2018-01-02 (Actual); Status verified 2017-12

CONDITIONS: Normal Tension Glaucoma; Bilirubin; Defect, Excretion
Keywords: serum bilirubin; normal-tension glaucoma; oxidative stress
MeSH Terms: conditions — Low Tension Glaucoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient group: This grup included 38 patients with NTG.
- Control group: This group included 38 healthy controls.

SUMMARY:
Purpose: To analyze the relationship between normal-tension glaucoma (NTG) and serum bilirubin levels.

Materials and Methods: This research included 38 patients with NTG and 38 healthy controls with similar age and sex distribution, for a total of 76 subjects. Serum samples were taken from all of the subjects, direct serum bilirubin, indirect serum bilirubin and the total serum bilirubin were measured.

DETAILED DESCRIPTION:
This is a retrospective study of cases with recently or previously diagnosed NTG who were admitted to our clinic between 2010 and 2017. This study included 38 patients with NTG and 38 healthy controls with similar age and sex distribution, for a total of 76 subjects. Written informed consent was obtained from all of the participants. The study was approved by the institutional review board of the hospital and adhered to the tenets of the Declaration of Helsinki.

A complete ophthalmic examination including best-corrected visual acuity, slit-lamp biomicroscopy, Goldmann applanation tonometry (AT 900, Haag-Streit Diagnostics, Koeniz, CH), corneal thickness evaluation (Pachymeter SP-3000, Tomey Corporation, Nagoya, JP), gonioscopy and ophthalmoscopy was performed in all NTG cases. Additionally, optical coherence tomography (OCT RS-3000 Lite, NIDEK Corporation, Tokyo, JP) measurement of the peripapillary retinal nerve fibre layer thickness, and Humprey visual field testing (Carl-Zeiss Meditec, Dublin, CA) were also performed.

NTG was diagnosed based on a clinical examination showing a normal IOP (corrected for corneal thickness), thinning of the peripapillary retinal nerve fibre layer, optic nerve damage, and characteristic glaucomatous visual field defects. The exclusion criteria included other forms of glaucoma such as primary open-angle glaucoma, primary closed-angle glaucoma, pigmentary glaucoma and exfoliative glaucoma. Patients who had active systemic diseases such as those affecting the liver, biliary system, pancreas and kidney and infectious diseases or malignant tumours that could influence the serum bilirubin concentrations were also excluded.

Fasting blood samples were taken from each participant to measure direct bilirubin, indirect bilirubin, and the total serum bilirubin concentrations. The direct bilirubin and total bilirubin concentrations were measured with an Architect C16000 Clinical Chemistry Analyzer (Abbott Laboratories, Abbott Park, IL, USA), using its original kits, and the indirect bilirubin concentrations were calculated by the following formula: indirect bilirubin = total bilirubin - direct bilirubin.

All the data were compiled into a computer file, and Statistical Package for Social Sciences for Windows 22.0 was used to perform the statistical analysis. Student's t test or the Mann-Whitney U test were used to compare the mean values between the two groups, after the evaluation of the data for a normal distribution using the Kolmogorov-Smirnov test. A p value less than 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* Patients who had active systemic diseases such as those affecting the liver, biliary system, pancreas and kidney and infectious diseases or malignant tumours that could influence the serum bilirubin concentrations were excluded.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: NTG was diagnosed based on a clinical examination showing a normal IOP (corrected for corneal thickness), thinning of the peripapillary retinal nerve fibre layer, optic nerve damage, and characteristic glaucomatous visual field defects. The exclusion criteria included other forms of glaucoma such as primary open-angle glaucoma, primary closed-angle glaucoma, pigmentary glaucoma and exfoliative glaucoma. Patients who had active systemic diseases such as those affecting the liver, biliary system, pancreas and kidney and infectious diseases or malignant tumours that could influence the serum bilirubin concentrations were also excluded.
Sampling Method: Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Serum Bilirubin Levels | January 2017-March 2017
  Serum indirect, direct and total bilirubin levels

CONTACTS AND LOCATIONS:
Overall Officials: Sadık Altan Ozal, Principal Investigator — Trakya University
Locations (1):
- Sadık Altan Ozal, Edirne, In the USA Or Canada, Please Select..., Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tham YC, Li X, Wong TY, Quigley HA, Aung T, Cheng CY. Global prevalence of glaucoma and projections of glaucoma burden through 2040: a systematic review and meta-analysis. Ophthalmology. 2014 Nov;121(11):2081-90. doi: 10.1016/j.ophtha.2014.05.013. Epub 2014 Jun 26. PMID 24974815
- [Result] Flammer J, Mozaffarieh M. What is the present pathogenetic concept of glaucomatous optic neuropathy? Surv Ophthalmol. 2007 Nov;52 Suppl 2:S162-73. doi: 10.1016/j.survophthal.2007.08.012. PMID 17998042
- [Result] Mallick J, Devi L, Malik PK, Mallick J. Update on Normal Tension Glaucoma. J Ophthalmic Vis Res. 2016 Apr-Jun;11(2):204-8. doi: 10.4103/2008-322X.183914. PMID 27413503
- [Result] Cho HK, Kee C. Population-based glaucoma prevalence studies in Asians. Surv Ophthalmol. 2014 Jul-Aug;59(4):434-47. doi: 10.1016/j.survophthal.2013.09.003. Epub 2014 May 13. PMID 24837853
- [Result] Iwase A, Suzuki Y, Araie M, Yamamoto T, Abe H, Shirato S, Kuwayama Y, Mishima HK, Shimizu H, Tomita G, Inoue Y, Kitazawa Y; Tajimi Study Group, Japan Glaucoma Society. The prevalence of primary open-angle glaucoma in Japanese: the Tajimi Study. Ophthalmology. 2004 Sep;111(9):1641-8. doi: 10.1016/j.ophtha.2004.03.029. PMID 15350316
- [Result] Cursiefen C, Wisse M, Cursiefen S, Junemann A, Martus P, Korth M. Migraine and tension headache in high-pressure and normal-pressure glaucoma. Am J Ophthalmol. 2000 Jan;129(1):102-4. doi: 10.1016/s0002-9394(99)00289-5. PMID 10653426
- [Result] Henry E, Newby DE, Webb DJ, O'Brien C. Peripheral endothelial dysfunction in normal pressure glaucoma. Invest Ophthalmol Vis Sci. 1999 Jul;40(8):1710-4. PMID 10393040
- [Result] Himori N, Kunikata H, Shiga Y, Omodaka K, Maruyama K, Takahashi H, Nakazawa T. The association between systemic oxidative stress and ocular blood flow in patients with normal-tension glaucoma. Graefes Arch Clin Exp Ophthalmol. 2016 Feb;254(2):333-41. doi: 10.1007/s00417-015-3203-z. Epub 2015 Oct 30. PMID 26514963
- [Result] Yuki K, Murat D, Kimura I, Ohtake Y, Tsubota K. Reduced-serum vitamin C and increased uric acid levels in normal-tension glaucoma. Graefes Arch Clin Exp Ophthalmol. 2010 Feb;248(2):243-8. doi: 10.1007/s00417-009-1183-6. Epub 2009 Sep 8. PMID 19763599
- [Result] Harada T, Harada C, Nakamura K, Quah HM, Okumura A, Namekata K, Saeki T, Aihara M, Yoshida H, Mitani A, Tanaka K. The potential role of glutamate transporters in the pathogenesis of normal tension glaucoma. J Clin Invest. 2007 Jul;117(7):1763-70. doi: 10.1172/JCI30178. PMID 17607354
- [Result] Gupta N, Singh T, Chaudhary R, Garg SK, Sandhu GS, Mittal V, Gupta R, Bodin R, Sule S. Bilirubin in coronary artery disease: Cytotoxic or protective? World J Gastrointest Pharmacol Ther. 2016 Nov 6;7(4):469-476. doi: 10.4292/wjgpt.v7.i4.469. PMID 27867680
- [Result] Kapitulnik J. Bilirubin: an endogenous product of heme degradation with both cytotoxic and cytoprotective properties. Mol Pharmacol. 2004 Oct;66(4):773-9. doi: 10.1124/mol.104.002832. Epub 2004 Jul 21. No abstract available. PMID 15269289
- [Result] Liao SL. The role of bilirubin and phototherapy in the oxidative/antioxidant balance. Pediatr Neonatol. 2015 Apr;56(2):77-8. doi: 10.1016/j.pedneo.2015.01.001. Epub 2015 Jan 22. No abstract available. PMID 25735960
- [Result] Wu TW, Fung KP, Wu J, Yang CC, Weisel RD. Antioxidation of human low density lipoprotein by unconjugated and conjugated bilirubins. Biochem Pharmacol. 1996 Mar 22;51(6):859-62. doi: 10.1016/0006-2952(95)02395-x. PMID 8602883
- [Result] Cao L, Xue L, Luo DM. Lower serum bilirubin concentration in patients with migraine. Int J Clin Exp Med. 2015 Aug 15;8(8):13398-402. eCollection 2015. PMID 26550273
- [Result] Vitek L, Jirsa M, Brodanova M, Kalab M, Marecek Z, Danzig V, Novotny L, Kotal P. Gilbert syndrome and ischemic heart disease: a protective effect of elevated bilirubin levels. Atherosclerosis. 2002 Feb;160(2):449-56. doi: 10.1016/s0021-9150(01)00601-3. PMID 11849670
- [Result] Peng F, Deng X, Yu Y, Chen X, Shen L, Zhong X, Qiu W, Jiang Y, Zhang J, Hu X. Serum bilirubin concentrations and multiple sclerosis. J Clin Neurosci. 2011 Oct;18(10):1355-9. doi: 10.1016/j.jocn.2011.02.023. Epub 2011 Jul 22. PMID 21782448
- [Result] Demir M, Demir C, Keceoglu S. Relationship between serum bilirubin concentration and nondipper hypertension. Int J Clin Exp Med. 2014 May 15;7(5):1454-8. eCollection 2014. PMID 24995111
- [Result] Tanindi A, Erkan AF, Alhan A, Tore HF. Arterial stiffness and central arterial wave reflection are associated with serum uric acid, total bilirubin, and neutrophil-to-lymphocyte ratio in patients with coronary artery disease. Anatol J Cardiol. 2015 May;15(5):396-403. doi: 10.5152/akd.2014.5447. Epub 2014 Jun 3. PMID 25430407